CLINICAL TRIAL: NCT06515353
Title: The Effect of Atmospheric Pressure on Patients Presenting to the Emergency Department With Gastrointestinal Bleeding
Brief Title: Gastrointestinal Bleeding and Atmospheric Pressure Relationship
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: GIB and Atmospheric Pressure
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Atmospheric Pressure; Adverse Effect; GastroIntestinal Bleeding
Keywords: atmospheric pressure; gastrointestinal bleeding; emergency department
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GI Bleeding: Patients administered to emergency department with GI bleeding will be scrrened and obtained retrospectively from hospital system.
  Atmospheric pressure data will be obtained from Meteorology Directorate. Patients' data will be evaluated according to atmospheric pressure values.

SUMMARY:
This study aims to investigate whether atmospheric pressure has an effect on upper gastrointestinal bleeding (UGIB), which includes causes such as peptic ulcer disease, esophagitis, gastritis, gastrointestinal varices, Mallory-Weiss tears, and gastric cancer. The goal is to determine the impact of atmospheric pressure and gather information on its role in high-risk UGIB.

DETAILED DESCRIPTION:
ur study aims to investigate the potential effects of changes in atmospheric pressure on gastrointestinal bleeding, and if such effects exist, to review treatment adjustments based on weather forecasts for hypertensive patients to prevent potential hypertensive emergencies and enhance patient comfort. This research poses no risk to patients and is purely observational and clinical in nature.

After initial evaluation upon presentation to the emergency department, patients will undergo routine emergency department monitoring for gastrointestinal bleeding, including physical examination, vital sign monitoring, evaluation of coagulation parameters, and hemoglobin levels. Apart from routine tests, no additional invasive or non-invasive procedures will be performed by us.

Obtained data from patients and atmospheric pressure data will be analyzed and evaluated. Results will be analyzed to determine any relation between gastrointestinal bleeding and atmospheric pressure changes

ELIGIBILITY:
Inclusion criteria:

Patients aged 18 and above Patients presenting to the emergency department with complaints of gastrointestinal bleeding, whether active or resolved Patients willing to participate in the study Patients from central districts of Ankara

Exclusion criteria:

Patients under the age of 18 Pregnant individuals Patients with a history of trauma at the time of admission Patients declaring they are from a city other than Ankara

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to emergency department with gastrointestinal bleeding
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
gastrointestinal bleeding | 24 hours
  patients administered to emergency department with gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo CG, Tian L, Zhang F, Cheung KS, Leung WK. Associations of seasonal variations and meteorological parameters with incidences of upper and lower gastrointestinal bleeding. J Gastroenterol Hepatol. 2021 Dec;36(12):3354-3362. doi: 10.1111/jgh.15632. Epub 2021 Jul 30. PMID 34289518
- [Background] Prechter F, Burger M, Lehmann T, Stallmach A, Schmidt C. A study on the correlation of gastrointestinal bleeding and meteorological factors - is there a weather condition for GI bleeding? Z Gastroenterol. 2019 Dec;57(12):1476-1480. doi: 10.1055/a-1008-9863. Epub 2019 Dec 11. PMID 31826278
- [Background] Lenzen H, Musmann E, Kottas M, Schonemeier B, Kohnlein T, Manns MP, Lankisch TO. Acute gastrointestinal bleeding cases presenting to the emergency department are associated with age, sex and seasonal and circadian factors. Eur J Gastroenterol Hepatol. 2017 Jan;29(1):78-83. doi: 10.1097/MEG.0000000000000752. PMID 27662496